CLINICAL TRIAL: NCT05069909
Title: Simplified Versus Conventional Complete Dentures: A Randomized Crossover Clinical Trial
Brief Title: Simplified Versus Conventional Complete Dentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Dr. Nadia Ereifej, AssociateProfessor, University of Jordan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: NEreifej
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Complete Edentulism
Keywords: Simplified dentures; impression techniques; complete edentulism; border moulding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional technique (Active Comparator): The group of patients who received dentures fabricated with conventional technique first
  Interventions: Procedure: Denture Fabrication technique
- Simplified technique (Active Comparator): The group of patients who received dentures fabricated with simplified technique first
  Interventions: Procedure: Denture Fabrication technique

INTERVENTIONS:
Procedure: Denture Fabrication technique — Each patient received two sets of dentures fabricated using the two different techniques and their satisfaction and OHIP-EDENT were compared

SUMMARY:
The purpose of this randomized, double-blind, 2-period crossover trial was to assess the satisfaction of edentulous patients and their oral health impact profile when provided with complete dentures fabricated using the conventional and simplified techniques.

DETAILED DESCRIPTION:
40 completely edentulous patients, aged 40-85 years, with no relevant medical conditions, seeking complete dentures at a university hospital were included in this study. Those were randomly divided into two groups (n=20). Each group received two sets of dentures, the Group (S) were given the dentures constructed using the simplified technique first while the Group (C) received the dentures constructed using the conventional technique. After 1 month of the first set of dentures delivery, participants were asked to rate their general satisfaction on a 10-cm visual analogue scale in addition to their satisfaction regarding comfort, retention, stability, efficiency of mastication and speaking. Participants were also asked to fill the 20-item oral health impact profile for edentulous patients (OHIP-EDENT). Thereafter, each group of patients were given the set of dentures constructed using the other technique, given instructions and recalled after 1 month to evaluate the alternate set of dentures. 2 Prosthodontists performed all the clinical procedures and 1 laboratory technician performed the laboratory procedures. The results of the study were analyzed using Wilcoxon-signed rank test at significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria

1. Patients seeking new conventional complete dentures for first time or as replacement of their previous complete dentures
2. Patients aged 40-85 y.
3. Patients who had been completely edentulous for at least 6 months
4. Patients who had well developed to moderately resorbed maxillary and mandibular ridges
5. Patients who had no denture fissuratum or any traumas from previous dentures
6. Patients who had no relevant medical issues, disorders of the masticatory system, neuromuscular dysfunction, auditory problems, psychological or psychiatric conditions that can affect the response to treatment, oral pathology, xerostomia, or tied tongue condition.
7. Patients had medical and dental insurance to cover the fees for construction of dentures by a Prosthodontic specialist
8. Patients who signed consent form

   -

   Exclusion Criteria:

   -

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction questionnaire | 1 month after denture delivery
  Visual analogue scale (0-10) for a 10 item questionnaire regarding patient satisfaction with the dentures
OHIP-EDENT | I month after denture delivery
  20-item oral health impact profile for edentulous patients questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol, Data analyses and results of both questionnaires will be shared